CLINICAL TRIAL: NCT05054751
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Clinical Trial of GB491 Combined With Fulvestrant in Subjects With HR+, HER2- Locally Advanced or Metastatic Breast Cancer Who Have Progressed on Prior Endocrine Therapy
Brief Title: GB491 Combined With Fulvestrant for HR+ HER2- Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GB491-004
Record Dates: First submitted 2021-08-13; First posted 2021-09-23 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
Keywords: CDK4/6; Phase III; GB491
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Evaluation; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB491+ Fulvestrant (Experimental)
  Interventions: Drug: GB491+ Fulvestrant
- Placebo+Fulvestrant (Placebo Comparator)
  Interventions: Drug: Placebo+Fulvestrant

INTERVENTIONS:
Drug: GB491+ Fulvestrant — GB491: The dose of GB491 is 150 mg, BID, which should be taken with a meal. The drug is administered according to the patient's dose group until the progression of disease or an intolerable toxicity occur or meet the criteria for termination of treatment or the patient withdraw informed consent or the sponsor discontinues the trial.
  Fulvestrant: Intramuscular injection of flurvexine 500mg on day 1 and day 15 of the first cycle, and flurvexine 500mg on day 1 of the second and subsequent cycles. Flurvexine 500mg should be given slowly (1-2 minutes per injection) on both sides of the buttocks, once 250 mg on each side. The drug is administered according to the patient's dose group until the progression of disease or an intolerable toxicity occur or meet the criteria for termination of treatment or the patient withdraw informed consent or the sponsor discontinues the trial.
  Other Names: test drug + Fulvestrant
  Arms: GB491+ Fulvestrant
Drug: Placebo+Fulvestrant — Placebo: The dose of Placebo is 150 mg, BID, which should be taken with a meal. The placebo is administered according to the patient's dose group until the progression of disease occur or meet the criteria for termination of treatment or the patient withdraw informed consent or the sponsor discontinues the trial.
  Fulvestrant: Intramuscular injection of flurvexine 500mg on day 1 and day 15 of the first cycle, and flurvexine 500mg on day 1 of the second and subsequent cycles. Flurvexine 500mg should be given slowly (1-2 minutes per injection) on both sides of the buttocks, once 250 mg on each side. The drug is administered according to the patient's dose group until the progression of disease or an intolerable toxicity occur or meet the criteria for termination of treatment or the patient withdraw informed consent or the sponsor discontinues the trial.
  Other Names: placebo control + Fulvestrant
  Arms: Placebo+Fulvestrant

SUMMARY:
GB491-004 is a multicenter, randomized, double-blind, placebo-controlled Phase III study to evaluate the efficacy and safety of GB491 in combination with fulvestrant in patients with HR-positive, HER2-negative locally advanced or metastatic breast cancer who have progressed on prior endocrine therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Females or males of 18 years of age or older and less than 75 years of age at study screening
2. Histologically or cytologically confirmed locally advanced or metastatic breast cancer that is not amenable to curative surgical resection or radiation therapy
3. Patients have been diagnosed with ER-positive breast cancer in the local laboratory
4. Patents have been diagnosed with HER2-negative breast cancer in the local laboratory
5. Menopausal status is not limited (including Premenopausal/perimenopausal/postmenopausal state)
6. Prior endocrine therapy and chemotherapy, the following are permitted:

1) Prior endocrine adjuvant therapy: a) Radiologic evidence of progressive disease (PD) during or within 12 months following (neo)adjuvant therapy with an aromatase inhibitor (AI) or an anti-estrogen such as tamoxifen, and no subsequent endocrine therapy for locally advanced or metastatic breast cancer; b) Radiologic evidence of PD during or within 12 months following (neo)adjuvant therapy with an AI or an anti-estrogen such as tamoxifen, after receiving the first-line endocrine therapy for locally advanced or metastatic breast cancer, and who developed radiologically documented PD after receiving therapy for ≥ 6 months; c) Radiologically documented PD more than 12 months following the end of adjuvant therapy with AIs or anti-estrogens such as tamoxifen, followed by radiographic progression following first-line therapy with AIs or anti-estrogens for locally advanced or metastatic breast cancer; 2) Progression with radiographic evidence of disease following prior first-line endocrine therapy for locally advanced or metastatic breast cancer in subjects who have not received prior (neo) adjuvant therapy; 3) Prior chemotherapy: In addition to endocrine therapy, subjects are eligible if they received a maximum of 1 prior line of chemotherapy for locally advanced or metastatic breast cancer and discontinued treatment for at least 28 days prior to randomization; 7.According to RECIST V1.1, the patient has at least one measurable lesion that has not been irradiated by radiotherapy and can be evaluated by CT/MRI; If there is no measurable lesion, there must be at least one osteolytic bone lesion that can be evaluated by CT/MRI 8.ECOG performance status of 0 or 1 9.Adequate organ and marrow function.

Key Exclusion Criteria:

1. Previous treatment with fulvestrant, everolimus or any other CDK4/6 inhibitors
2. Patients with known hypersensitivity to any component of GB491 or Fulvestrant
3. Known active, uncontrolled, or symptomatic central nervous system metastasis, carcinomatous meningitis, or clinically manifested leptomeningeal disease, cerebral edema, spinal compression or/and tumor progressive growth
4. Visceral crisis
5. Patients with skin lesion only and radiographically non-measurable at baseline
6. Persistent toxicities (CTCAE Grade >2) caused by previous anticancer therapy, excluding alopecia
7. Patients who have been on bisphosphonates and denosumab therapy at a stable dose for less than 7 days prior to randomization
8. Patients who have received limited field radiotherapy in 2 weeks or extended field radiotherapy in 4 weeks before randomization or radiation with more than 30% of the bone marrow
9. Patients use drugs or fruits containing strong inducers or inhibitors of CYP3A4/5, or drugs with narrow therapeutic window that are mainly metabolized by CYP3A4/5 in 14 days before randomization
10. Patients with long-term systematic use of corticosteroids
11. Any severe and/or uncontrollable medical conditions
12. Patients with severely impaired lung function
13. Known history of HIV infection or history of HIV seropositivity
14. Patients have significant hepatic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
PFS assessed by the investigator | Approximately 1.5 years
  To assess the PFS assessed by the investigator

SECONDARY OUTCOMES:
PFS assessed by the blinded independent central review (BICR) | Approximately 1.5 years
  To assess the PFS assessed by the BICR
OS | Approximately 3 years
  To assess the overall survival (OS)
ORR | Approximately 1.5 years
  To assess the objective response rate (ORR)
DOR | Approximately 1.5 years
  To assess the duration of response
DCR | Approximately 1.5 years
  To assess the disease control rate
CBR | Approximately 1.5 years
  To assess the clinical benefit rate
Safety and tolerability | Approximately 3 years
  To assess the safety and tolerability assessed by incidence and severity of adverse events (AEs) and serious AEs (SAEs) according to NCI-CTCAE version 5.0
PK | From Cycle 1 to Cycle 4, approximately 4 months
  To assess the PK assessed by population pharmacokinetic analysis based on plasma concentrations of GB491

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (54):
- China (54):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chaoyang Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Cancer hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital , Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chognqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First people's hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong provincial TCM hospital, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences,Shenzhen Center Shenzhen Cancer Hospital, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Hainan Third People's Hospital, Sanya, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated hospital of Hebei University, Shijiazhuang, Hebei
  - Harbin Medcial Univercity cancer hospital, Haerbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Affiliated hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Bethune First Hospital Of Jilin University, Changchun, Jillin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer hospital & Institute, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated hospital of Jining Medical University, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The first hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China School of Medicine, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Third Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu B, Zhang Q, Luo Y, Tong Z, Sun T, Shan C, Liu X, Yao Y, Zhao B, Wang S, Zeng X, Hu C, Yan X, Wang X, Jia H, Chen Z, Qiu F, Wu X, Zhang D, Li T. Lerociclib plus fulvestrant in patients with HR+/HER2- locally advanced or metastatic breast cancer who have progressed on prior endocrine therapy: LEONARDA-1 a phase III randomized trial. Nat Commun. 2025 Jan 16;16(1):716. doi: 10.1038/s41467-025-56096-2. PMID 39820749